CLINICAL TRIAL: NCT06995989
Title: Combined Effects of Energy Conservation Techniques With Pursed Lip Breathing on Functional Independence and Quality of Life in Bronchiectasis
Brief Title: Effects of Energy Conservation Techniques With Pursed Lip Breathing on Quality of Life in Bronchiectasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0358
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis, breathing exercises , Dyspnea
MeSH Terms: conditions — Bronchiectasis; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- energy conservation techniques along with pursed lip breathing technique (Experimental): Group A will receive energy conservation techniques with pursed lip breathing with
  1 session a day for total 5 days in a week. 1 session will consist of 3 cycles of pursed lip breathing for duration of 10 minutes with a break of 20 minutes in between. ECTs will be trained for 2 weeks. A detailed manual will be developed to ensure the consistency of the training for all subjects. Examples of interventions are training to use ergonomic principles along with pursed lip breathing. The subjects were trained to place their equipment at chest height; they were trained to work at paced speed and in some cases instructed to use technical aids.
  Interventions: Other: energy conservation techniques with pursed lip breathing
- pursed lip breathing technique (Experimental): Group B will receive pursed lip breathing
  Interventions: Other: pursed lip breathing

INTERVENTIONS:
Other: energy conservation techniques with pursed lip breathing — Group A will receive energy conservation techniques with pursed lip breathing with
  1 session a day for total 5 days in a week. 1 session will consist of 3 cycles of pursed lip breathing for duration of 10 minutes with a break of 20 minutes in between. ECTs will be trained for 2 weeks. A detailed manual will be developed to ensure the consistency of the training for all subjects. Examples of interventions are training to use ergonomic principles along with pursed lip breathing. The subjects were trained to place their equipment at chest height; they were trained to work at paced speed and in some cases instructed to use technical aids.
  Arms: energy conservation techniques along with pursed lip breathing technique
Other: pursed lip breathing — pursed lip breathing
  Arms: pursed lip breathing technique

SUMMARY:
Bronchiectasis is the abnormal dilatation of the bronchi. Due to airway dilatation patient is unable to clear the mucus and risk of infection is increased. For mucus clearance used many breathing techniques employed along with or without mechanical devices. Many researches have shown the inconsistent results of energy conservation techniques along with breathing exercises among variety of cardiopulmonary disorders. This study will be conducted to determine the combined effects of energy conservation techniques with pursed lip breathing on functional independence and quality of life in patients of bronchiectasis. It will be a randomized clinical trial. Two groups will be taken under the age of 40 to 60 years and data will be collected from pulmonary wards of selected hospitals. Sample size will be 46 keeping the attrition rate 10%.

St. George's Respiratory Questionnaire (SGRQ) will be used to evaluate the quality of life of patients and 6 mint walk test is used to determine functional independence of bronchiectasis patients. After data collection, data will be analyzed using SPSS version 26.

DETAILED DESCRIPTION:
Bronchiectasis is the abnormal dilatation of the bronchi. Due to airway dilatation patient is unable to clear the mucus and risk of infection is increased. For mucus clearance and reduced labored breathing, conventional chest physiotherapy is used in which many breathing techniques can be employed along with or without mechanical devices and inspiratory muscle training, coughing support and positioning to improve the respiratory functions but there is no consensus on which breathing technique is better. Many researches have shown the inconsistent results of energy conservation techniques along with breathing exercises among variety of cardiopulmonary disorders such as in asthma, chronic obstructive pulmonary disease (COPD) patients but no results were seen among patients of bronchiectasis. This study will be conducted to determine the combined effects of energy conservation techniques with pursed lip breathing on functional independence and quality of life in patients of bronchiectasis. It will be a randomized clinical trial. Age of selected subjects will be between 40 to 60 years and data will be collected from pulmonary wards of selected hospitals. Sample size will be 46 keeping the attrition rate 10%. There will be 2 groups i.e. group A will receive energy conservation techniques along with pursed lip breathing technique and group B will receive only pursed lip breathing technique. St. George's Respiratory Questionnaire (SGRQ) will be used to evaluate the quality of life of patients and 6 mint walk test is used to determine functional independence of bronchiectasis patients. After data collection, data will be analyzed using SPSS version 26.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, aged between 40 to 60 years Bronchiectasis

Exclusion Criteria:

* Prior history of open-heart surgery

  * Prior severe pulmonary/hepatic or renal disease
  * Life-threatening arrhythmias (ventricular fibrillation, ventricular tachycardia, atrial fibrillation)
  * Pulmonary complications (atelectasis, acute respiratory distress syndrome (ARDS), diaphragmatic injury)
  * Congestive heart failure
  * Deep venous thrombosis (DVT)
  * Any known psychological disease

Ages: 40 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-05-28 (Estimated); Primary Completion 2025-09-28 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
St. George's Respiratory Questionnaire (SGRQ) | 2 weeks
  Patients completed on paper the SGRQ, it includes dimensions for SGRQ activity, SGRQ impact, SGRQ symptoms, and SGRQ total. The scale ranges from 0 (excellent quality of life) to 100 (worst quality of life) for all four dimensions
6 Minutes walk test | 2 weeks
  The patient is asked to walk as far as possible along a 30-m minimally trafficked corridor for a period of 6 min with the primary outcome measure being the 6-min walk distance (6MWD) measured in meters

CONTACTS AND LOCATIONS:
Overall Officials: Arjumand Bano, MS-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Sadiq hospital Sargodha, DHQ Sargodha, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No